CLINICAL TRIAL: NCT02087007
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel Group, Therapeutic Confirmatory Study to Evaluate the Efficacy and Safety of Pletaal(Cilostazol) in Subjects With Vasospastic Angina
Brief Title: A Therapeutic Confirmatory Study to Evaluate the Efficacy and Safety of Cilostazol in Subjects With Vasospastic Angina
Acronym: STELLA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Korea Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 021-KOA-1301i
Record Dates: First submitted 2014-02-17; First posted 2014-03-14 (Estimated); Last update posted 2017-05-04 (Actual); Status verified 2017-05

CONDITIONS: Vasospastic Angina
Keywords: Treatment for vasospastic angina
MeSH Terms: conditions — Angina Pectoris, Variant | interventions — Cilostazol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- group 1 (Experimental): Cilostazol 50mg, Cilostzaol 100mg
  Interventions: Drug: Cilostazol
- group 2 (Placebo Comparator): placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Cilostazol — 100mg oral tablets bid during 2 weeks after dosing of 50mg oral tablets bid during 2 weeks
  Arms: group 1
Drug: placebo — 100mg oral placebo tablets bid during 2 weeks after dosing of 50mg oral placebo tablets bid during 2 weeks
  Arms: group 2

SUMMARY:
This study will be conducted in accordance with the local regulation of New Drug Application. Overall duration of this trial will be 3 years after approval of KFDA.

Each subject will participate around 7 weeks, which include the 2 weeks Amlodipine run-in period, 4 weeks double blind period and 1 week safety follow up period

DETAILED DESCRIPTION:
A Multicenter, Randomized, Double-Blind, Placebo-controlled, Parallel group, Therapeutic confirmatory Study.

The subject who has at least one episode of chest pain weekly and at least two episodes of chest pain during last week despite Amlodipine 5mg qd taking during 2 weeks will have treatment of Pletaal(Cilostazol) or Placebo for 4 weeks. Pletaal(Cilostazol) is taken 100mg oral tablets bid during 2 weeks after dosing of Pletaal(Cilostazol) 50mg oral tablets bid during 2 weeks. Placebo of Pletaal(Cilostazol) is used as the control medication.

ELIGIBILITY:
Subjects must meet all of the following inclusion criteria to be eligible for enrollment into the study :

1. Male or female 20 or over the age of 20 and under the age of 80.
2. Patients showing angina attack even while resting during the screening, diagnosed with vasospastic angina within the previous 3 months by meeting at least one of the 3 definitions, and accompanying insignificant (stenosis rate <50%) coronary artery disease documented by coronary angiography within the last 3 months [temporary antispastic agents (monotherapies or a combination of Verapamil and Nitroglycerin, anticoagulants) for coronary angiography are allowed]

   * Chest pain accompanied by at least 2 temporary, closely located ST elevations or depressions of 0.1mV or greater in the absence of ergonovine provoked coronary angiography.
   * Positive Intracoronary (IC) or Intravenous (IV) Ergonovine provocation test; ischemic ECG change accompanied by chest pain and spasm reducing the coronary diameter by 90% or more (at least 2 temporary, closely located ST elevations or depressions of 0.1mV or greater on 12-lead ECG)
3. Patients who reported at least 1 episode of chest pain in a week during amlodipine run-in period and at least 2 episodes in the final week.
4. Women who had been menopausal or sterile for at least 1 year, or women of childbearing potential who agree to practice a contraceptive measure throughout the clinical trial (e.g., hormonal contraceptives, intrauterine devices, condom + spermicidal agents, diaphragm + spermicidal agents, and partner's infertility)
5. Subjects who signed a written agreement indicating that they were given full explanations of the clinical trial and are willing to participate in the clinical trial.

Subjects presenting with any of the following will not be included in the study:

1. Subjects who used Cilostazol within 3 months before the screening visit
2. Subjects who used antiplatelet drugs, including Aspirin, Clopidogrel, Ticlopidine and Sarpogrelate, or PDE3 inhibitors of the same class as Cilostazol, such as Amrinone, Milrinone and Enoximone, after the initiation of the amlodipine run-in period
3. Subjects who used oral anticoagulants, such as warfarin, within 1 months prior to the screening visit
4. Subjects who used any of the following drugs within 1 week prior to the screening visit

   * CCBs apart from amlodipine
   * Beta-blockers or alpha-blockers
   * Oral nitrate, excluding nitroglycerin sublingual tablet, Nicorandil
   * Vitamin E preparations
   * Estrogens
5. History of myocardial infarction or with myocardial infarction mediated by vasospastic angina at the time of screening
6. History of a life-threatening vasospastic event (e.g., ventricular tachycardia, atrial fibrillation or syncope)
7. History of stroke, intracranial hemorrhage or transient ischemic attack (TIA)
8. Hemorrhage (hemophilia, capillary fragility, upper gastrointestinal bleeding, urinary tract bleeding, hemoptysis, vitreous hemorrhage, etc.) or such predisposition (active peptic ulcer, hemorrhage suspected at Cilostazol administration for surgical wound within the last 3 months, proliferative diabetic retinopathy)
9. History of hypersensitivity to the ingredients of Cilostazol, amlodipine, dihydropyridines such as nitroglycerine, and nitrates
10. Severe aortic stenosis
11. History of shock
12. Hypotension with systolic pressure of below 90mmHg at screening
13. Severe anemia with hemoglobin 6.5g/dl or below at screening
14. History of glaucoma
15. ST change abnormality not interpretable on ECG at screening
16. Congestive heart failure with left ventricular ejection fraction <40% on echocardiography at screening or within the last 3 months
17. Atrial fibrillation or beyond moderate valvular heart disease
18. Left main coronary spasm suspected or confirmed by coronary angiography or ergonovine provoked coronary angiography
19. History of coronary artery bypass graft (CABG) or percutaneous coronary intervention (PCI)
20. Heart rate >100 bpm at screening via vital sign: tachycardia
21. Uncontrolled hypertension with systolic pressure ≥ 160 mmHg or diastolic pressure ≥ 100 mmHg at screening
22. Creatinine level ≥ 1.5 mg/dL at screening
23. AST or ALT > x3 ULN(Upper Limit of Normal) at screening
24. Platelet count < 100,000mm3 at screening
25. QT prolongation of QTcB > 450 msec in male and QTcB>470 msec in female subjects at screening
26. Women of childbearing potential with positive pregnancy test at screening
27. Women who did not agree to practice a contraceptive measure, pregnant or lactating women
28. Drug compliance of less than 80% during 2-week amlodipine run-in period
29. Subjects otherwise judged by the investigator to be inappropriate for inclusion in the trial
30. Subjects who used another investigational products within 2 months prior to the randomization

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2013-11; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Chest Pain Frequency | Baseline and Week 4
  Change of the chest pain frequency on the final a week after IP dosing from a week before IP dosing

SECONDARY OUTCOMES:
Percent change of the chest pain frequency | Baseline and Week 4
  Percent change of the chest pain frequency on the final a week after IP dosing from a week before IP dosing
Proportion of subjects without chest pain | 4 weeks
  Proportion of subjects without chest pain on the final a week after IP dosing
total chest pain intensity | Baseline and Week 4
  Change of the total pain intensity on the final a week after IP dosing from a week before IP dosing
average pain intensity(the total pain intensity/the number of pain) | Baseline and Week 4
  Change of the average pain intensity(the total pain intensity/the number of pain) on the final a week after IP dosing from a week before IP dosing
total nitroglycerin sublingual consumption | Baseline and Week 4
  Change of the total nitroglycerin sublingual consumption of the final a week after IP dosing from a week before IP dosing

CONTACTS AND LOCATIONS:
Locations (1):
- Yangsan Busan University Hospital, Busan, South Korea